CLINICAL TRIAL: NCT02316119
Title: Mechanisms Involved in the Bleeding Risk of Patients With Coronary Artery Diseased Previous Stroke or Transient Ischemic Attack in Use of Antiplatelet Therapy
Brief Title: Mechanistic Study of Bleeding Risk in Coronary Patients With Cerebrovascular Disease
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: FAPESP2012/04930-0
Record Dates: First submitted 2014-12-03; First posted 2014-12-12 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Artery Disease; Cerebral Stroke; TIA (Transient Ischemic Attack)
Keywords: bleeding risk, acute coronary syndrome, platelet agregation,
MeSH Terms: conditions — Coronary Artery Disease; Stroke; Ischemic Attack, Transient; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Post-ACS patients without history of IS/TIA previously to the acute coronary and taking aspirin
- Case group: Post ACS patients with history of IS/TIA previously to the acute coronary event and taking aspirin

SUMMARY:
Background: About 5% of patients with acute coronary syndrome (ACS) have had previously ischemic stroke (IS) or transitory ischemic attack (TIA). This is a high-risk population, with a high incidence of ischemic events, and also of bleeding events. While the high ischemic risk in this population is attributed to a higher prevalence of cardiovascular risk factors, their predisposition to bleeding events is not well understood. Hypothesis: The increased bleeding risk in ACS patients with history of cerebrovascular event may be justified by a low platelet activity. Methods: Unicentric, prospective, case-control study, which included approximately 100 post-ACS patients with history of IS/TIA previously to the acute coronary event (Case Group) and 100 patients without IS/TIA (Control group). The groups were matched for gender, age, and ACS type and year of occurrence. All patients were taking aspirin, and the main exclusion criteria were use of dual antiplatelet therapy, previous hemorrhagic stroke, severe renal dysfunction, thrombocytopenia or coagulopathy. Main analysis: Platelet aggregation was evaluated by 6 methods: VerifyNow Aspirin®, VerifyNow P2Y12®, PFA 100®, thrombelastography (ReoRox®), light transmission aggregometry with ADP (LTA ADP) and epinephrine (LTA EPI) as agonists. Additional analysis: genetic, HDL transport and inflammatory evaliation

ELIGIBILITY:
Inclusion Criteria:

* Post-ACS patients with history of IS/TIA previously to the acute coronary event and taking aspirin
* Sign the consent form

Exclusion Criteria:

* Hemorrhagic stroke
* Another antiplatelet drug than aspirin
* Use of Anti inflammatory drug
* Severe chronic kidney dysfunction
* Liver disease
* Coagulopathy
* Platelet disfunction
* Thrombocytopenia or thrombocytosis
* Refuse to sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-ACS patients and taking aspirin
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Residual platelet activity by VerifyNow Aspirin (Aspirin reactivity units) | in the selection visit

SECONDARY OUTCOMES:
Baseline platelet activity by VerifyNow P2Y12 (P2Y12 reactivity units) | in the selection visit

OTHER OUTCOMES:
light transmission aggregometry with ADP (maximum amplitude) | in the selection visit
light transmission aggregometry with epinephrine (maximum amplitude) | in the selection visit
platelet acitivity by PFA 100® (seconds) | in the selection visit
kinetics of clot by thromboelastography usin Reorox ® (seconds, paschal/min, paschal) | in the selection visit

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical unit of acute coronary disease, São Paulo, São Paulo, Brazil